CLINICAL TRIAL: NCT05535257
Title: Pilot Study to Establish Use of Lower Extremity Sleeve and Sequential Compression Pump Device in Patients With Upper Extremity Weakness Post-Stroke
Brief Title: A Study to Evaluate Lower Extremity Sleeve and Pump Device to Treat Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Suzanne K. Langley, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-009068
Record Dates: First submitted 2022-08-19; First posted 2022-09-10 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Upper Extremity Weakness; Stroke
MeSH Terms: conditions — Paresis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Sequential Compression Device (SCD) on upper extremity (Experimental): Subjects post stroke with upper extremity weakness have the SCD sleeve placed on the arm for up to 4 hours for one day only
  Interventions: Device: Sequential Compression Device

INTERVENTIONS:
Device: Sequential Compression Device — Calf size lower extremity sequential compression device sleeve will be placed on the weak upper extremity blow the cubital fossa and may include the hand if necessary. The device will inflate and deflate.
  Other Names: SCD

SUMMARY:
The primary purpose of this study is to establish that application of a Sequential Compression Device (SCD) and lower extremity (LE) sleeve applied to a hemi-paretic upper extremity is safe.

DETAILED DESCRIPTION:
Studies has shown that passively stimulating the arm with vibration can improve sensory and motor recovery and movement. Researchers want to expand on this with a more advanced stimulation but in a device that is already routinely used. The SCD is normally used to prevent blood clots. It uses pressure to keep blood moving in the leg. It is routinely used in hospitals across the country. While it does this it warms and even vibrates the leg giving many types of stimulation to the limb and to the brain. This stimulation may help improve recovery further, at marginal cost, while possibly reducing the chances of blood clots in an immobile limb.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Mayo Clinic/Jacksonville, post-stroke with a hemiparetic upper extremity.
* Able to provide consent of participation by self-agreement.
* Patients with a hemiparetic upper extremity will be determined using the NIH Motor Arm subsection from the NIH scale and score a 1-4.
* Patients who have received thrombolytic therapeutic medicine > 13 hours (per site specific policy) will not be excluded from inclusion in this study.
* Patients who score > 13 on the BIMS to ensure intact cognition.

Exclusion Criteria:

* Inability to provide consent of participation.
* Subjects with aphasia or the inability to effectively communicate their pain consistently.
* Questionable reliability scoring < 13 on the BIMS, has an existing invasive line (PICC line, IV, AV fistula or AV graft); recent surgery or vein ligation in the involved extremity.
* Recent skin graft in the involved extremity.
* Confirmed DVT in the affected.
* Upper extremity including axillary or subclavian veins; open or active wounds or infection in the involved extremity.
* Upper extremity ischemia, gangrene, cellulitis or severe arteriosclerosis in the affected upper extremity.
* Status-post axillary lymph node dissection on the involved side; congestive heart failure (CHF) acute exacerbation; acute edema of unknown etiology in the involved upper extremity.
* Subjects with extreme deformity of the affected upper extremity.
* Subjects with an acute kidney injury.
* Subjects who are hemodynamically unstable 1,7,17.
* Patients who have received thrombolytic therapeutic medicine administered < 13 hours (per site specific policy) prior to application of SCD sleeve.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Langley, OT, Principal Investigator — Mayo Clinic
Locations (1):
- C Joseph Yelvington, Saint Johns, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period for 20 subjects enrolled in this study was from 9/27/2022 to 11/14/2023. All subjects were recruited and enrolled in the Mayo Clinic Hospital setting.
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: Subjects post stroke with upper extremity weakness and impaired sensation have the SCD sleeve placed on the arm for up to 4 hours for one day only
  Sequential Compression Device: Calf size lower extremity sequential compression device sleeve will be placed on the weak upper extremity blow the cubital fossa and may include the hand if necessary. The device will inflate and deflate.
Period: Overall Study
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: Subjects post stroke with upper extremity weakness had the SCD sleeve placed on the arm for up to 4 hours for one day only Device: Sequential Compression Device Calf size lower extremity sequential compression device sleeve was placed on the weak upper extremity blow the cubital fossa and may include the hand if necessary. The device inflated and deflated,
  Other Names:
  SCD
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Wearing Tolerance of the SCD and Sleeve on the Upper Extremity.
Description: Number of subjects who answered yes to the question "Are you tolerating this sleeve"
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: Wearing tolerance outcome measure results of 20 subjects based on 4 hour wearing trial
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Pain With SCD Sleeve and Device
Description: Total number of subjects to report No pain measured by Visual Analogue Scale (VAS) where patient identifies pain on a line between "no pain" and "worst possible pain".
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: Pain outcome measure on 20 subjects
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
Number analyzed (Participants) | 20
Participants | 20

3. Other Pre Specified Outcome: Nail Bed Color
Description: Nail bed color will be observed and described/documented with terms of "normal", "dusky", or "bluish" in color
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: Nail bed color (normal, blue, dusky)
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
Number analyzed (Participants) | 20
Participants
  Normal | 20
  Bluish | 0
  Dusky | 0

4. Other Pre Specified Outcome: Edema Measured in Inches of Circumference of Forearm
Description: Using tape measure the weak UE forearm will be measured in inches; 5 inches distal to cubital fossa, proximal from the wrist crease.
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: Edema on UE forearm upper 2/3 below cubital fossa
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
Number analyzed (Participants) | 20
Participants
  1.5 inch decrease in circumference | 2
  1.25 inch decrease in circumference | 2
  1 inch decrease in circumference | 2
  .5 inch decrease in circumference | 1
  .25 inch decrease in circumference | 6
  No change in circumference | 3
  .25 inch increase in circumference | 4

5. Other Pre Specified Outcome: UE Strength Using Motor Arm Subsection #5 of NIH Scale
Description: The limb is placed in the appropriate position: extend the arm (palm down) 90 degrees if sitting or 45 degrees if supine. Drift is scored if the arm falls before 10 seconds. Documenting using Scale definition: 0=No drift, 1=Drift, 2=Some effort against gravity, 3=No effort against gravity; limb falls, 4=No movement
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: UE Strength using Motor Arm subsection #5 of NIH scale
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
Number analyzed (Participants) | 20
Participants
  4 (no movement) | 2
  3 (no effort against gravity) | 3
  2 (some effort against gravity) | 5
  1 (drift) | 8
  0 (no drift) | 2

6. Other Pre Specified Outcome: UE Sensation
Description: Using cotton swab and lightly touching skin at dermatome points C2, C3, C4, C5, C6, C7, C8, T1, T2 using the International Standards for the Classification of Spinal Cord Injury Key Sensory Points documenting "Intact" or "Impaired"
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: UE Sensation
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
Number analyzed (Participants) | 20
Participants
  Sensation Intact | 10
  Sensation Impaired | 10

7. Other Pre Specified Outcome: UE Skin Integrity
Description: Prior to placement of sleeve and upon removal of sleeve during check time skin will be visually assessed and the terms "Intact" or "Impaired" will be documented. Any new "redness", "rash", or "bruising" and "area" of arm will be documented and the need to remove sleeve at that time will be determined.
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: UE Skin Integrity
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
Number analyzed (Participants) | 20
Participants
  Intact Skin Integrity | 20
  Impaired Skin Integrity | 0

8. Other Pre Specified Outcome: UE Grip Strength
Description: Using dynamometer in pounds measures affected hand strength at baseline and at 4-hours for each subject. This outcome measure was added approximately 1/2 way through the subject recruitment as a revision to this study to help capture subjects with hand weakness who may not have gross arm weakness (captured by Motor arm Subsection #5 outcome measure).
Time Frame: Baseline and at four-hours for each subject
Measure: Count of Participants; unit: Participants
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: UE hand/grip strength measured in pounds using dynamometer to affected hand only
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
Number analyzed (Participants) | 11
Participants
  0 lbs baseline and 0 at 4 hours | 5
  30 lbs at baseline and 34 lbs at 4 hours | 1
  12 lbs at baseline and 10 lbs at 4 hours | 1
  65 lbs at baseline and 62 lbs at 4 hours | 1
  35 lbs at baseline and 35 lbs at 4 hours | 1
  20 lbs at baseline and 2 lbs at 4 hours | 1
  32 lbs at baseline and 38 lbs at 4 hours | 1

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected during the wearing trial (4 hours) of each subjects participation from dates 9/27/2022 to 11/14/2023
Groups:
- Sequential Compression Device (SCD) on Upper Extremity: Stroke patients with UE weakness and or sensory impairments.
Arm/Group | Sequential Compression Device (SCD) on Upper Extremity
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT05535257/Prot_000.pdf